CLINICAL TRIAL: NCT01017666
Title: A Randomized, Double-Blind, Placebo-Controlled, Crossover Study to Assess the Effect of BIIB014 on the Pharmacokinetics of Rosiglitazone, Warfarin, and Midazolam in Healthy Volunteers
Brief Title: BIIB014 Effects on the Pharmacokinetics (PK) of Rosiglitazone, Warfarin, and Midazolam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 204HV103; EUDRA CT 2009-014259-60
Record Dates: First submitted 2009-11-16; First posted 2009-11-20 (Estimated); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Healthy
Keywords: Healthy Volunteer
MeSH Terms: interventions — 3-(4-amino-3-methylbenzyl)-7-(2-furyl)-3H-(1,2,3)triazolo(4,5-d)pyrimidine-5-amine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rosiglitazone 8mg PO (Experimental): Cohort 1
  Interventions: Drug: BIIB014; Drug: Placebo
- Midazolam 2mg PO, Warfarin 25mg PO (Experimental): Cohort 2
  Interventions: Drug: BIIB014; Drug: Placebo

INTERVENTIONS:
Drug: BIIB014 — BIIB014 100mg PO Cohort 1 - 8d Cohort 2 - 14d
Drug: Placebo — Matched placebo to BIIB014 Cohort 1 - 8d Cohort 2 - 14d

SUMMARY:
The purpose of this study is to understand whether BIIB014 has potential to affect how certain drugs are broken down by the body.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects
* Between the ages of 18 and 45, inclusive.
* Must have a body mass index (BMI) between 19 kg/m2 and 30 kg/m2, inclusive

Exclusion Criteria:

* Clinically significant abnormalities (as determined by the Investigator)
* Other unspecified reason that would make the subject unsuitable for enrollment (as determined by the Investigator)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2009-11-01 (Actual); Primary Completion 2010-06-02 (Actual); Study Completion 2010-06-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile of rosiglitazone (Cohort 1), midazolam & metabolites and s-warfarin (Cohort 2) during steady state exposure to BIIB014 or placebo | 24 hours (Cohort 1); 144 hours (Cohort 2)

SECONDARY OUTCOMES:
Adverse Events | Duration of subject participation

CONTACTS AND LOCATIONS:
Locations (1):
- InCROM Clinical Research Unit, London, United Kingdom